CLINICAL TRIAL: NCT06484920
Title: A Phase II Study of the Combination of Pembrolizumab and All-Trans Retinoic Acid Combination Treatment of Relapsed Hodgkin Lymphoma (HL) and B-Non-Hodgkin- Lymphoma (B-NHL)
Brief Title: A Phase II Study of the Combination of Pembrolizumab and ATRA Combination Treatment of Relapsed HL and B-NHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rita Assi (Other)
Responsible Party: Sponsor-Investigator, Rita Assi, Assistant Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0866
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Relapsed Hodgkin Lymphoma; Refractory Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; B-cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATRA and Pembrolizumab (Experimental): Patients will receive 200mg Q3W pembrolizumab treatment plus the supplemental treatment of 150 mg/m2 ATRA orally for 3 days surrounding each of the first four infusions of pembrolizumab (day -1, day 0, day +1).
  Interventions: Drug: ATRA; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ATRA — 150 mg/m2 ATRA orally for 3 days surrounding each of the first four cycles (day -1, day 0, day +1)
Drug: Pembrolizumab — 200mg Q3W pembrolizumab

SUMMARY:
This is a Phase II single-center open label trial of the combination of ATRA and pembrolizumab treatment in patients with histologically proven, relapsed or refractory Hodgkin Lymphoma or B-Non-Hodgkin-lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Willingness to comply with all study procedures and be available for the duration of the trial
4. Have a performance status of 0 to 2 on the ECOG Performance Scale.
5. Life expectancy ≥12 weeks as per investigator discretion
6. Patients with histologically proven, relapsed or refractory HL or B-NHL as follows:

   1. HL after failure of at least 1 prior line of systemic therapy
   2. Primary mediastinal large B-cell lymphoma (PMBCL) that is refractory to first-line therapy
   3. Other B-cell NHLs after failure of at least 2 prior lines of systemic therapy. The eligible types of B-cell NHLs are:

   i. Diffuse large B cell lymphoma ii. Follicular lymphoma iii. Marginal Zone lymphoma iv. Mantle Cell Lymphoma d. Indolent lymphoma are only eligible if they require systemic treatment e. Lymphocyte predominant HL are eligible Note: Formalin-fixed, paraffin embedded archival tumor sample from the primary cancer must be available for testing. If not available or sufficient, patients will be asked to undergo an US or CT guided biopsy prior to study entry to satisfy this eligibility criterion.
7. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 10 days prior to the first study treatment: Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) INR and aPTT ≤1.5 x ULN; this applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose. Renal calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) calculated creatinine clearance ≥ 60 mL/min Hepatic Serum total bilirubin

   * 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN (patients with known Gilbert disease who have bilirubin levels ≤ 3 x ULN may be enrolled). Patients must be able to undergo biliary stenting if required before or, if required, during the trial AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR
   * 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: Female of childbearing potential definition: (ECOG definition) Any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

   1. Has not undergone a hysterectomy or bilateral oophorectomy; or
   2. Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
9. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.

   Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

   Refer to section 8.4.1 for more information.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception of the protocol, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Refer to section 8.4.1 for more information.
11. Acceptable methods of contraception include IUD, oral contraceptive, subdermal implant, and double barrier (condom with a contraceptive sponge or contraceptive pessary). Micro-dosed progesterone preparations ("mini-pill") are an inadequate method of contraception during treatment with ATRA. If patients are taking this pill they should be instructed to stop, and another form of contraceptive should be prescribed instead.
12. Patients with a history of CAR-T cell therapy are eligible if ≥ 3 months post treatment.

Exclusion Criteria:

1. Patients currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Known brain metastases and/or leptomeningeal disease. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
3. Significant reduction in ECOG performance status between the screening/ baseline visit and within 72 hours prior to commencement of treatment as per trial protocol, as per the Investigator's assessment, defined as a reduction in ECOG score to 3 or 4.
4. Patients with a diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) within 7 days prior to the first dose of trial treatment.

   Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Contraindication to the use of ATRA including but not limited to: patients with a history of hypersensitivity reaction to tretinoin, vesanoid or related compounds ( i.e. acitretin, isotretinoin, vitamin A); , Tetracyclines, Progesterone (low dose), drugs inducing P450 (rifampicin, glucocorticoids, phenobarbital, etc), ketoconazole and drugs inhibiting p450 (cimetidine, erythromycin, cyclosporine, etc); antifibrinolytic agents (e.g. tranexamic acid, aminocaproic acid, aprotinin) and hydroxyurea)
7. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day -1 or who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. Prior chemotherapy targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day -1 or who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Subjects with chronic conditions such as vision changes or prior hearing loss that is not reasonably expected to be exacerbated by the investigational product may be included. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: Subjects with Grade 2 adrenal insufficiency or thyroid conditions who are not expected to resolve to baseline, are on a stable dose of medication may be included if it is not reasonably expected to be exacerbated by the investigational product, and asymptomatic whilst on treatment.
9. History of malignancy in the last 5 years with the exception of prior history of in situ cancer or basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
10. Patient has undergone major surgery, other than diagnostic surgery (i.e., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day -1 of treatment in this study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
11. Known history of, or any evidence of active, non-infectious pneumonitis.
12. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
13. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
16. Patients on micro-dosed progesterone preparations ("mini-pill") who are unwilling to receive an alternative form of contraception.
17. Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
18. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
19. Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
20. known history of active TB (Bacillus Tuberculosis).
21. Receipt of live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
22. Patients who receive a COVID shot and/or booster within 4 weeks of Cycle 1 Day -1.
23. Known sensitivity to retinoic acid derivatives.
24. Patient is taking any prohibited concurrent medication, including Vitamin A supplements, and CYP3A modulators (inducers and inhibitors) and is unwilling to stop use (washout period of 3 days for this protocol) prior to treatment start and during the trial.
25. History of allogenic stem cell transplant or received a solid organ transplant. Note: If history of transplant is ≥ 5 years, subjects may be deemed eligible at the discretion of the treating physician. Note: Patients with a history of autologous stem cell transplant performed for lymphoma are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | from start of treatment through 90 days safety follow-up visit
  Safety will be assess by the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Overall Response Rate | Screening to up to 2 years post last therapy
Complete Remission Rate | Screening to up to 2 years post last therapy
Patient derived myeloid-derived suppressor cells (MDSC) | Screening, before cycle 2, before cycle 4, and within 60 days after cycle 4 day 1
  Assessing the anti-tumor effect of the combination of pembrolizumab and ATRA on the reduction in myeloid-derived suppressor cells (MDSC) frequency and suppressive function through in vitro experiments using patient-derived MDSCs.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Assi, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Health Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided